CLINICAL TRIAL: NCT03744273
Title: Capsule Biopsy in Acellular Dermal Matrix-based Prosthetic Breast Reconstruction: a Prospective Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jai-Kyong Pyon, Professor, Principal Investigator, Samsung Medical Center
Other Study IDs: 2012-03-028
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasms; Mammaplasty; Acellular Dermis
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

INTERVENTIONS:
Procedure: breast capsule biopsy

SUMMARY:
In this prospective study, breast capsule biopsy was performed in patients undergoing 2-stage expander-implant breast reconstruction to determine its use. Prospective clinical trial was designed for 10 consecutive patients as a pilot study and approved by IRB of Samsung Medical Center. From November 2013 to May 2015, full-thickness capsule biopsy specimen was obtained from acellular dermal matrix (ADM) capsule and from native subpectoral capsule (internal control) during expander-implant exchange. Biopsy specimens were scored for fibrosis and inflammatory reactions.

This is completed study and its specific title, study objective, method, and results will be available online after scientific journal submission.

ELIGIBILITY:
Inclusion Criteria:

* age between 20 and 70
* planning 2-stage expander-implant breast reconstruction using acellular dermal matrix
* with no medical history such as diabetes, hypertension, or smoking
* no surgical history

Exclusion Criteria:

* pregnant
* newly detected medical or surgical condition
* acellular dermal matrix loss due to allergic reaction or prosthetic infection
* breast cancer recurrence
* transfer to other institution
* reconstruction give-up due to patient's wish
* no biopsy score

Ages: 20 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2013-11-03 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2015-05-26 (Actual)

PRIMARY OUTCOMES:
histology scoring | immediate after biopsy
  semiquantitative histopathologic score system of biopsy specimens (reference: Basu et al., Plastic and Reconstructive Surgery, 126: 1842, 2010)

CONTACTS AND LOCATIONS:
Overall Officials: Jai-Kyong Pyon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea